CLINICAL TRIAL: NCT00565383
Title: The Effect of Combined Spinal-Epidural Analgesia on the Success of External Cephalic Version for Breech Position
Brief Title: The Effect of Combined Spinal-Epidural Analgesia on the Success of External Cephalic Version (ECV) for Breech Position
Acronym: Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Sullivan, John T. Sullivan M.D., Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0897-002; Sullivan 002 (Other: NorthwesternU)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Pregnancy; Breech Presentation
Keywords: Pregnancy; 37 Weeks Gestation; Breech Presentation; Version Procedure; Pain Control; Neuraxial analgesia
MeSH Terms: conditions — Breech Presentation; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous fentanyl analgesia (Active Comparator): Intravenous fentanyl (50 mcg) analgesia
  Interventions: Procedure: Intravenous fentanyl (50mcg)
- Combined spinal-epidural analgesia (Experimental): Combined spinal-epidural analgesia (intrathecal fentanyl 2.5 mg plus bupivacaine 2.5 mg) single administration
  Interventions: Procedure: Combined spinal-epidural analgesia

INTERVENTIONS:
Procedure: Combined spinal-epidural analgesia — Combined spinal-epidural
  Arms: Combined spinal-epidural analgesia
Procedure: Intravenous fentanyl (50mcg) — Intravenous fentanyl
  Arms: Intravenous fentanyl analgesia

SUMMARY:
We aim to answer the clinical question: Does combined spinal-epidural analgesia improve the success rate of external cephalic version? We hypothesize that neuraxial analgesia (spinal or epidural analgesia) during version for breech presentation increases successful fetal rotation and decreases the incidence of Cesarean delivery for malpresentation.

DETAILED DESCRIPTION:
At term 2 to 3% of singleton pregnancies are in breech presentation. Many of these deliveries are managed by cesarean delivery due to higher neonatal morbidity associated with vaginal breech delivery. Cesarean delivery, the safer option for the baby, however, is associated with a higher incidence of maternal complications for both the current and subsequent pregnancies. External cephalic version is a procedure commonly used to attempt to manually rotate the fetus into vertex position. This facilitates vaginal delivery and thus avoids higher maternal and/or neonatal complications.

Obstetricians perform versions after 36 weeks gestational age with a reportable success rate of 30-80%. The most common technique involves external manipulation of the fetal position preceded by pharmacologic uterine relaxation. Pain relief is most commonly provided in the form of intravenous opioids such as fentanyl. A more efficacious form of analgesia is the use of neuraxial opioids and local anesthetics (neuraxial analgesia), a technique commonly used for labor and delivery analgesia.

Although the use of neuraxial analgesia and anesthesia techniques improve maternal pain and satisfaction, there is conflicting evidence if they improve the success rate of version procedures. The American College of Obstetricians and Gynecologists (ACOG) has stated, "Currently there is not enough evidence to make a recommendation favoring or opposing anesthesia during ECV (external cephalic version) attempts."

We propose to conduct a prospective, single blinded, randomized clinical trial to assess the impact of combined spinal-epidural analgesia on the success rate of external version for breech fetal position and the subsequent incidence of vaginal vs. Cesarean delivery as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Female
* Pregnant
* Breech Presentation
* Greater than 36 Weeks gestation
* Version Procedure

Exclusion Criteria:

* Under 18 or over 55 years of age

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2002-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Does combined spinal-epidural analgesia improve the success rate of external cephalic version? | Time between analgesia intervention for the version procedure and delivery

SECONDARY OUTCOMES:
Mode of delivery | At delivery
Maternal satisfaction | Between analgesic intervention and the completion of the version procedure
Maternal Pain | Between analgesic intervention and termination of the version procedure

CONTACTS AND LOCATIONS:
Overall Officials: John T Sullivan, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Fortunato SJ, Mercer LJ, Guzick DS. External cephalic version with tocolysis: factors associated with success. Obstet Gynecol. 1988 Jul;72(1):59-62. PMID 3288930
- [Background] Zhang J, Bowes WA Jr, Fortney JA. Efficacy of external cephalic version: a review. Obstet Gynecol. 1993 Aug;82(2):306-12. PMID 8336883
- [Background] Carlan SJ, Dent JM, Huckaby T, Whittington EC, Shaefer D. The effect of epidural anesthesia on safety and success of external cephalic version at term. Anesth Analg. 1994 Sep;79(3):525-8. doi: 10.1213/00000539-199409000-00021. PMID 8067558
- [Background] Birnbach DJ, Matut J, Stein DJ, Campagnuolo J, Drimbarean C, Grunebaum A, Kuroda MM, Thys DM. The effect of intrathecal analgesia on the success of external cephalic version. Anesth Analg. 2001 Aug;93(2):410-3, 4th contents page. doi: 10.1097/00000539-200108000-00035. PMID 11473871